CLINICAL TRIAL: NCT00047801
Title: Phase 1-2a Dose-Ranging Study of TLK286 in Combination With Docetaxel (Taxotere) in Platinum-Resistant Non-Small Cell Lung Cancer
Brief Title: Phase 1-2a Dose-Ranging Study of TLK286 in Combination With Docetaxel in Platinum-Resistant Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Telik (Industry)
Responsible Party: Gail Brown, M.D. Chief Medical Officer, Telik, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TLK286.2012; NCT00068705 (obsolete NCT alias)
Record Dates: First submitted 2002-10-18; First posted 2002-10-21 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-06

CONDITIONS: Carcinoma, Non-small-cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — TER 286; Docetaxel

INTERVENTIONS:
Drug: TLK286 in combination with docetaxel

SUMMARY:
The purpose of this study is to determine the effectiveness and safety of TLK286 given intravenously once every three weeks in combination with docetaxel (Taxotere) in the treatment of patients with non-small cell lung cancer that is resistant to platinum-based chemotherapy.

ELIGIBILITY:
Inclusion criteria include:

* Histologically confirmed non-small cell bronchogenic carcinoma, including squamous cell carcinoma, undifferentiated carcinoma, adenocarcinoma, mixed (adenocarcinoma with squamous cell carcinoma), bronchoalveolar carcinoma, or large cell carcinoma
* Stage IV or Stage IIIB
* Progressed during or after first-line therapies with platinum-containing regimens in the advanced or metastatic treatment regimen
* At least 18 years of age
* Good performance status (ECOG 0 to 1)
* Adequate liver, renal, and bone marrow function

Exclusion criteria include:

* Pregnant or lactating women
* Treatment with more than one cytotoxic therapy
* Prior radiation to the whole pelvis
* Unstable medical conditions such as uncontrolled cardiac arrhythmia
* Patients with known history of severe hypersensitivity reactions to docetaxel or other drugs formulated with polysorbate 80

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28
Dates: Start 2002-10; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Cancer Institute Medical Group, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Indiana University Cancer Center, Indianapolis, Indiana
  - M.D. Anderson Cancer Center, Houston, Texas